CLINICAL TRIAL: NCT05934903
Title: Feasibility Study: tDCS for Treatment of Refractory Status Epilepticus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet adequate enrolment numbers for feasibility.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 2000035450; No NIH funding (Other: 10.11.23)
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Status Epilepticus; Refractory Status Epilepticus
Keywords: Transcranial Direct Current Stimulation; Ictal-Interictal Continuum; Neurostimulation; Seizures; Epilepsy
MeSH Terms: conditions — Status Epilepticus; Seizures; Epilepsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double blind block randomized into stimulation arm versus sham stimulation arm.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will not know the treatment arm, and the outcomes assessor reading electroencephalogram will not know treatment arm. The device does not have a sham mode so study personnel applying the device will be aware of the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation (Experimental): The tDCS device will stimulate with a 2mA current during sessions. Both arms receive application of the device for 3 sessions of 2x 30 minute active application with 30 minutes rest in between.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Stimulation (Sham Comparator): The tDCS device will stimulate with a 0mA current during sessions (sham). Both arms receive application of the device for 3 sessions of 2x 30 minute active application with 30 minutes rest in between.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Cathodal direct current stimulation at 0 or 2mA will be applied to subjects

SUMMARY:
Status epilepticus, or recurrent seizures without return to baseline, is a neurologic emergency. Refractory status epilepticus occurs when seizures are resistant to multiple first line anti-seizure medications. The ability to quickly stop seizures is paramount. Transcranial direct current simulation is a non-invasive, easily administered therapy that can potentially help reduce seizure burden.

The goal of this feasibility study is to assess the ability of the study site to enroll patients admitted with refractory seizures or those with abnormal brain wave patterns to take part in a study looking to use transcranial direct current stimulation as an adjunctive treatment. The main questions it aims to answer are:

* What is the recruitment capability of the study site?
* How well can the study site adhere to study protocol?
* Are there any adverse effects of using the transcranial direct current stimulation device?
* How do patients' brain wave studies respond to the stimulation? Participants will be asked to consider joining the study. Once joined, researchers will randomly assign participants to compare transcranial stimulation versus sham stimulation to see if this will affect the participant's brain wave patterns.

DETAILED DESCRIPTION:
This is study is designed to determine the feasibility of implementing a double-blinded tDCS in inpatients with status epilepticus and other abnormal EEG (electroencephalography) patterns. The study includes assessments of recruitment capability, the ability to implement the study procedures, the safety profile, and preliminary evaluation of participant response to transcranial direct current stimulation (tDCS) therapy, to see which clinical outcome measures are most practical.

Patients who are admitted to Yale New Haven Hospital with refractory status epilepticus or EEG patterns falling on the ictal-interictal continuum (IIC, rhythmic or periodic patterns with rates more than 1Hz and less than or equal to 2.5Hz) will be recruited, starting from August 1st 2023 until July 31st 2025, or until 60 total participants, whichever is sooner. Those who are eligible will be randomized into two groups: stimulation or sham, all while receiving standard of care according to their primary teams.

Each subject will receive up to 3 sessions of tDCS over a 72 hour period with at least 24 hours between each session. Each session will consist of 30 minutes of stimulation (or sham), a 30 minute break and a second 30 minute of stimulation (or sham). Stimulation will be applied using the ActivaDose II device (Caputron). Saline soaked sponges will be prepared, with the cathode being placed on the area corresponding to the seizure focus or point of maximal epileptic potential as defined on the international 10-20 EEG system. The anode will be placed on the contralateral shoulder. During each session, a maximum of total injected current across the electrodes of 2mA will be used, as conventional tDCS with 2mA is well-tolerated in adults and children. Sham stimulation includes application of the electrodes and timing the device to deliver 0mA of injected current.

The patients will not be aware of their randomization arm. The research staff analyzing the EEG data will not be aware of the patient's treatment arm.

The study schedule will include:

1. Screening and Consent visit
2. Stimulation Sessions - 3 one-hour stimulation sessions, distributed over 72 consecutive hours, and no less than 24 hours apart.
3. Follow up visit at 30 days after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient with refractory status epilepticus (RSE), or supra-refractory status epilepticus (SRSE), or electroencephalographic (EEG) characteristics > 50% of the time on the ictal-interictal continuum (IIC) or epilepsia partialis continua for at least 12 hours.

  * A patient with RSE is defined as having seizure(s) refractory to first line benzodiazepines and second-line antiseizure medications (ASMs; phenytoin, levetiracetam, valproate).
  * A patient with SRSE is defined as:

    * requiring at least 24 hours of a third-line intravenous anesthetic therapy (IVAT) such as propofol, midazolam, or ketamine, and
    * failing at least one previous wean of an IVAT.
  * A patient with epilepsia partialis continua (EPC) is defined as:

    * having focal seizure(s) refractory to first line benzodiazepines and second-line ASMs and
    * repeated episodes lasting more than one hour
  * A patient on the IIC is defined as:

    * having periodic discharges or rhythmic patterns at a rate at more than 1Hz and less than 3Hz and
    * IIC patterns for more than 50% of the time (IIC burden = 50%) within any prior 12 hour interval.
* access to continuous EEG monitoring
* brain imaging (Computerized Tomography or Magnetic Resonance Imaging) within 1 year of presentation

Exclusion Criteria:

* Damaged skin on scalp as determined by the primary team that prevents reasonably accurate electroencephalography monitoring and which may interfere with tDCS stimulation.
* Cranial metal implants (>1 mm thick epicranial titanium skull plates and metal dental fillings) or medical devices (i.e. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant).
* Previous surgeries opening the skull leaving skull defects capable of allowing the insertion of a cylinder with a radius greater or equal to 5 mm.
* Presence of any disease, medical condition or physical condition that, in the opinion of the Investigators, may adversely impact the safety of the subject or the integrity of the data
* Those who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment capability of the study site- Incidence | up to 24 months
  Recruitment capability of the study site will be assessed as the incidence of patients admitted with RSE/SRSE or IIC burden > 50% within a 24 month period. Participants admitted undergoing cEEG monitoring will be screened for having RSE or IIC burden >50% on a weekly basis.
Recruitment capability of the study site- Prevalence | up to 24 months
  Recruitment capability of the study site will be assessed as the prevalence of patients admitted with RSE/SRSE or IIC burden > 50% within a 24 month period. Participants admitted undergoing cEEG monitoring will be screened for having RSE or IIC burden >50% on a weekly basis.
  Prevalence will be calculated against weekly average patient census.
Recruitment capability of the study site- Percent Eligible | up to 24 months
  Recruitment capability of the study site will be assessed as the percent of eligible study participants compared to all patients admitted with RSE or IIC burden >50% within a 24-month period.
Recruitment capability of the study site- Percent Consent | up to 24 months
  Recruitment capability of the study site will be assessed as the percent of eligible participants who consent for study
Recruitment capability of the study site- Percent Withdraw | up to 24 months
  Recruitment capability of the study site will be assessed as the percent of consented participants who withdraw consent.

SECONDARY OUTCOMES:
Ability to implement protocol at study site | up to 24 months
  Ability to implement protocol at the study site will be assessed as the percent of patients able to complete the stimulation protocol and drop out causes.
Ability to implement protocol at study site- Protocol Deviations | up to 24 months
  Ability to implement protocol at the study site will be assessed as the percent of protocol deviations including un-blinding, contamination, truncation or extension of stimulation protocol, and qualitative causes of protocol deviations.
Ability to implement protocol at study site- Participants Lost to Follow Up | up to 24 months
  Ability to implement protocol at the study site will be assessed as the percent of participants lost to follow up.
Ability to implement protocol at study site- Device Failures | up to 24 months
  Ability to implement protocol at the study site will be assessed as the percent of device failure compared to total number of stimulation sessions.
Safety profile of tDCS by number of adverse events. | up to 24 months
  Safety profile of tDCS will be assessed as the number of adverse events.
Safety profile of tDCS by number of serious adverse events. | up to 24 months
  Safety profile of tDCS will be assessed as the number of serious adverse events.
Preliminary evaluation of effect of tDCS- Change in Time to resolution of status epilepticus | Baseline, 12 hours, 24 hours, 7 days, and 30 days
  Preliminary evaluation of the effect of tDCS on participants with RSE/SRSE or high IIC burden will be assessed as time to resolution of status epilepticus in patients admitted with RSE and SRSE (hours) in either study arm. Time to resolution of status epilepticus is defined as the time from first stimulation session until cessation of electrographic status epilepticus for more than 8 hours.
Preliminary evaluation of effect of tDCS- Change in Seizure Burden | Baseline, 12 hours, 24 hours, 7 days, and 30 days
  Preliminary evaluation of the effect of tDCS on participants with RSE/SRSE or high IIC burden will be assessed using EEG assessments to determine seizure burden before, during, and after intervention. Assesments will be conducted by study personnel on a post-hoc basis and quantified using both automatic spike detection software (Persyst) and manual methods.
Preliminary evaluation of effect of tDCS- Change in IIC burden | Baseline, 12 hours, 24 hours, 7 days, and 30 days
  Preliminary evaluation of the effect of tDCS on participants with RSE/SRSE or high IIC burden will be assessed using EEG assessments to determine IIC burden before, during, and after intervention. Assessments will be conducted by study personnel on a post-hoc basis and quantified using both automatic spike detection software (Persyst) and manual methods.
Preliminary evaluation of effect of tDCS- Change in ASM burden | Baseline, 12 hours, 24 hours, 7 days, and 30 days
  Preliminary evaluation of the effect of tDCS on participants with RSE/SRSE or high IIC burden will be assessed by the ASM burden at baseline, 12 hours, 7 days, and 30 days after intervention. Anti-seizure medication burden is defined as the sum total of all antiseizure medication ratios. Antiseizure medication ratios are defined as the prescribed total daily dose given over the maximal allowed daily dose of each given antiseizure medication as defined by the World Health Organization as the typical daily dose for a given ASM. ASM burden = Σ (ASM total daily dose/ASM total daily max dose).
Preliminary evaluation of effect of tDCS- Change in Acute Physiology and Chronic Health Evaluation (APACHE) II Score | Baseline and 7 days
  Preliminary evaluation of the effect of tDCS on participants with RSE/SRSE or high IIC burden will be assessed using the APACHE II Score. Each variable is weighted from 0 to 4, with the range of the total score from 0 to 71. Higher scores correspond to more severe disease and a higher risk of death.
Preliminary evaluation of effect of tDCS- Change in modified Rankin Score | Baseline and 30 days
  Preliminary evaluation of the effect of tDCS on participants with RSE/SRSE or high IIC burden will be assessed using the modified Rankin Score. It is a 6 point disability scale with possible scores ranging from 0 (no disability) to 5.(disability requiring constant care for all needs); 6 is death.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Quraishi, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trinka E, Rainer LJ, Granbichler CA, Zimmermann G, Leitinger M. Mortality, and life expectancy in Epilepsy and Status epilepticus-current trends and future aspects. Front Epidemiol. 2023 Feb 23;3:1081757. doi: 10.3389/fepid.2023.1081757. eCollection 2023. PMID 38455899
- [Background] Fisher RS, McGinn RJ, Von Stein EL, Wu TQ, Qing KY, Fogarty A, Razavi B, Venkatasubramanian C. Transcranial direct current stimulation for focal status epilepticus or lateralized periodic discharges in four patients in a critical care setting. Epilepsia. 2023 Apr;64(4):875-887. doi: 10.1111/epi.17514. Epub 2023 Feb 7. PMID 36661376
- [Background] Ng MC, El-Alawi H, Toutant D, Choi EH, Wright N, Khanam M, Paunovic B, Ko JH. A Pilot Study of High-Definition Transcranial Direct Current Stimulation in Refractory Status Epilepticus: The SURESTEP Trial. Neurotherapeutics. 2023 Jan;20(1):181-194. doi: 10.1007/s13311-022-01317-5. Epub 2022 Nov 2. PMID 36323975
- [Background] Matsumoto H, Ugawa Y. Adverse events of tDCS and tACS: A review. Clin Neurophysiol Pract. 2016 Dec 21;2:19-25. doi: 10.1016/j.cnp.2016.12.003. eCollection 2017. PMID 30214966
- [Background] Yang D, Wang Q, Xu C, Fang F, Fan J, Li L, Du Q, Zhang R, Wang Y, Lin Y, Huang Z, Wang H, Chen C, Xu Q, Wang Y, Zhang Y, Zhang Z, Zhao X, Zhao X, Li T, Liu C, Niu Y, Zhou Q, Zhou Q, Duan Y, Liu X, Yu T, Xue Q, Li J, Dai X, Han J, Ren C, Xu H, Li N, Zhang J, Xu N, Yang K, Wang Y. Transcranial direct current stimulation reduces seizure frequency in patients with refractory focal epilepsy: A randomized, double-blind, sham-controlled, and three-arm parallel multicenter study. Brain Stimul. 2020 Jan-Feb;13(1):109-116. doi: 10.1016/j.brs.2019.09.006. Epub 2019 Sep 24. PMID 31606448